CLINICAL TRIAL: NCT05587218
Title: How Motor Cortex Supports L2 Acquisition of Spoken Words, Signs, and Characters Via Perception and Production
Brief Title: Recognition of Second Language Spoken Words, Signs, and Characters Via Perception and Production in Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: L2WordProd
Record Dates: First submitted 2022-09-30; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-09

CONDITIONS: Second Language Acquisition in Healthy Young Adults
Keywords: Second language; Word learning; Self-production

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-production (Experimental): L2 lexical items self-produced at learning
  Interventions: Behavioral: Self-production
- Perception (Active Comparator): L2 lexical items heard or observed an additional time at learning
  Interventions: Behavioral: Self-production

INTERVENTIONS:
Behavioral: Self-production — After participants learn L2 lexical items via hearing or observing them paired with L1 translations, they are prompted to produce them themselves

SUMMARY:
Self-production facilitates acquisition of spoken words, signs, and characters from an unfamiliar second language. The proposed work investigates how motor cortex, a key part of the brain enabling body action, supports their acquisition via production as well as perception, providing insight into whether they are learned via mental simulation of the body actions used to produce them. It is hypothesized that activity in motor cortex will differ based on the body part used to produce lexical items (e.g., mouth vs. hands), will be greater for lexical items learned via production than observation, and will differentiate lexical items recognized successfully vs. unsuccessfully.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Native English speaker

Exclusion Criteria:

* Knowledge of sign language or languages with logographic characters
* Hearing or vision impairments
* Speech, language, or learning disorders
* Unsecured metal body implants

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-23 (Estimated); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
Functional activity in motor cortex location, 5 min, recognition | 5 minutes after learning
  Location of Blood Oxygen Level Dependent (BOLD) signal in motor cortex at recognition
Functional activity in motor cortex degree, 5 min, recognition | 5 minutes after learning
  Degree of Blood Oxygen Level Dependent (BOLD) signal in motor cortex at recognition
Functional activity in motor cortex location, 1 week, recognition | 1 week after learning
  Location of Blood Oxygen Level Dependent (BOLD) signal in motor cortex at recognition
Functional activity in motor cortex degree, 1 week, recognition | 1 week after learning
  Degree of Blood Oxygen Level Dependent (BOLD) signal in motor cortex at recognition

CONTACTS AND LOCATIONS:
Overall Officials: Laura Morett, Ph.D., Principal Investigator — University of Alabama, Tuscaloosa
Locations (1):
- University of Alabama, Tuscaloosa, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) underlying results in publications (de-identified)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately upon publication
Access Criteria: Publicly available